CLINICAL TRIAL: NCT02382809
Title: Efficacy of DC071 Mouthwash (0.2% Chlorhexidine Digluconate) in Peri-surgical Care for Preventing Alveolar Osteitis After Third Molar Extraction
Brief Title: Efficacy of 0.2 % Digluconate Chlorhexidine Mouthwash for Preventing Alveolar Osteitis After Third Molar Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DC0071 BB 4 05; 2014-004682-24 (EudraCT Number)
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Alveolar Osteitis
Keywords: Alveolar osteitis; Third molar; Dry socket; Mouthwash; third molar extraction
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- DC071 (0.2% chlorhexidine digluconate) (Experimental)
  Interventions: Drug: DC071
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DC071 — Mouthwash, twice daily
  Arms: DC071 (0.2% chlorhexidine digluconate)
Drug: Placebo — Mouthwash, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy of 0.2 % digluconate chlorhexidine mouthwash in the prevention of alveolar osteitis following third molar extraction and to evaluate the safety and local tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 years old
* Subject needing to undergo extraction of one impacted mandibular third molar
* For woman of childbearing potential and woman in post menopausal period under hormonal substitution treatment, she must accept to plan the extraction of the impacted mandibular third molar only during the last week of the menstrual cycle.
* Affiliated to a social security system, or is a beneficiary (if applicable in the national regulation)

Exclusion Criteria:

* Existence or history of parotid gland disorders
* Acute or history of recent acute pericoronitis at any tooth
* Extraction of more than 1 third molar in the same surgical procedure
* Subject at high risk of bacterial endocarditis (prosthetic heart valve, history of bacterial endocarditis, congenital cyanogenic heart disease)
* Coagulation or haemostatic disorder or use of anticoagulants
* Hypersensitivity to chlorhexidine or any of the excipients;
* Hypersensitivity to any anesthetic agent;
* Hypersensitivity to corticosteroids, analgesics including opioid drugs used for post-surgery pain relief
* Intake of systemic vasodilator or vasoconstrictor
* Intake of systemic or local (in the mouth) antibiotics within 7 days before Day 1 and/or any pre- or post-operative antibiotic prophylaxis planned to be prescribed during the study;
* Use of any antiseptic mouthwash within 7 days before Day -1
* Regular heavy smokers (more than 20 cigarettes per day)
* Is pregnant or in post-partum period or a nursing mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of an alveolar osteitis | Within 7 days
  The primary Outcome measure will be evaluated based on the absence/presence of an alveolar osteitis within 7 days after the extraction of the third molar.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise TONNER, Study Director — Pierre Fabre Medicament
Locations (18):
- Tallinn, Estonia
- France (10):
  - Bordeaux
  - Brest
  - Dijon
  - Le Petit-Quevilly
  - Lyon
  - Metz
  - Pierre-Bénite
  - Saint-Maixent-l'École
  - Strasbourg
  - Toulouse
- Latvia (4):
  - Daugavpils
  - Liepāja
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius